CLINICAL TRIAL: NCT00404443
Title: Efficacy of Traditional Chinese Acupuncture in the Treatment of Rheumatoid Arthritis: a Double-Blind Controlled Pilot Study
Brief Title: Acupuncture for the Treatment of Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Lai-Shan Tam, The Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCM04001
Record Dates: First submitted 2006-11-27; First posted 2006-11-28 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Acupuncture; Electroacupuncture; Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Sham Comparator): arm 1: placebo needle
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — Placebo-needles 17 will be used for those randomized to receive sham-acupuncture, which will be connected to the electrical current generator for the same duration and at the same acupuncture points without any current passing through, and intermittent non-specific manual twirling will also be applied. Patients are discouraged to communicate with each other before and after the treatment sessions to minimize bias.

SUMMARY:
To study the efficacy of acupuncture used as an adjunct measure for patients with refractory RA

DETAILED DESCRIPTION:
The study employs a randomized, prospective, double-blind, placebo-controlled trial to evaluate the effect of electroacupuncture, traditional Chinese acupuncture and sham acupuncture in patients with refractory RA. All patients received 20 sessions over a period of 10 weeks. Six acupuncture points were chosen. Primary outcome is the changes in the pain score. Secondary outcomes included the changes in the ACR core disease measures, DAS 28 score and the number of patients who achieved ACR 20 at week 10.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilled The American College of Rheumatology (ACR)[10] criteria of RA
* Active disease affecting the hands and wrists defined as having at least 4 tender joints and 2 swollen joints
* Early morning stiffness of greater than 45 minutes
* ESR > 28 mmHg or CRP > 10
* Patients taking disease modifying anti-rheumatic drugs (DMARDs) were eligible if they were on a stable dose for at least 3 months before screening.
* Patients on stable doses of one non-steroidal anti-inflammatory drug (NSAID) or up to 10 mg daily prednisone were also included.

Exclusion Criteria:

* Under the age of 18 years
* Pregnancy
* Previously had acupuncture
* Localized skin infections
* Anticoagulated
* Bleeding diathesis
* Intra-articular corticosteroid within 4 weeks preceding the study
* Any severe chronic or uncontrolled co-morbid disease
* Fear of needles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-12; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
The changes in the pain score. | wk52

SECONDARY OUTCOMES:
The ACR core disease measures | wk52
DAS 28 score | wk52
The number of patients who achieved ACR 20 at week 10. | wk52

CONTACTS AND LOCATIONS:
Overall Officials: Edmund K Li, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Institute of Chinese Medicine, Hong Kong, China

REFERENCES:
- [Derived] Tam LS, Leung PC, Li TK, Zhang L, Li EK. Acupuncture in the treatment of rheumatoid arthritis: a double-blind controlled pilot study. BMC Complement Altern Med. 2007 Nov 3;7:35. doi: 10.1186/1472-6882-7-35. PMID 17980044